CLINICAL TRIAL: NCT01726894
Title: A Prospective Development Study Evaluating Focal Therapy Using Irreversible Electroporation (Nanoknife®) in Men With Localised Prostate Cancer
Brief Title: Focal Therapy for Localised Prostate Cancer Using Irreversible Electroporation
Acronym: Nano
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Professor Mark Emberton, Professor, University College London Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 12/0399
Record Dates: First submitted 2012-10-30; First posted 2012-11-15 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer
Keywords: Focal Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irreversible Electroporation (Experimental)
  Interventions: Device: Irreversible Electroporation

INTERVENTIONS:
Device: Irreversible Electroporation

SUMMARY:
To determine the adverse events and genito-urinary side-effect profile of focal therapy to treat localised low to intermediate risk prostate cancer using irreversible electroporation (Nanoknife™).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer, Gleason Score </=7
* An anterior visible lesion on mpMRI, that is accessible to IRE treatment
* Transperineal prostate biopsies (template mapping and/or limited targeted) correlating with clinically significant lesion in the area of the MR-visible lesion (within 2 Barzell zones)
* Absence of clinically significant disease outside of the planned treatment zone, from histopathology and/or mpMRI findings
* Stage radiologicalT1-T2cN0M0 disease, as determined by local guidelines
* Serum PSA </=15 ng/ml
* Life expectancy of >/= 10 years
* Signed informed consent by patient
* An understanding of the English language sufficient to understand written and verbal information about the trial and consent process

Exclusion Criteria:

* Men who have had previous radiation therapy
* Men who have had androgen suppression/hormone treatment within the previous 12 months for their prostate cancer
* Men with evidence of metastatic disease or nodal disease outside the prostate on bone scan or cross-sectional imaging
* Men with a non-visible tumour on mpMRI
* Men with an inability to tolerate a transrectal ultrasound
* Men with latex allergies
* Men who have undergone prior significant rectal surgery preventing insertion of the TRUS probe (decided on the type of surgery in individual cases)
* Men who have had previous IRE, HIFU, cryosurgery, thermal or microwave therapy to the prostate.
* Men who have undergone a Transurethral Resection of the Prostate (TURP) for symptomatic lower urinary tract symptoms within 6 months. These patients may be included within the trial if deferred from consenting and screening until at least 6 months following the TURP.
* Men not fit for major surgery as assessed by a Consultant Anaesthetist
* Men unable to have pelvic MRI scanning (severe claustrophobia, permanent cardiac pacemaker, metallic implant etc likely to contribute significant artefact to images)
* Presence of metal implants/stents in the urethra
* Men with renal impairment with a GFR of <35ml/min (unable to tolerate Gadolinium dynamic contrast enhanced MRI).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Safety Profile | Up to 1 year
  Number of patients with adverse events using the National Cancer Institute Common Terminology Criteria (NCI CTC) classification system.

SECONDARY OUTCOMES:
Sexual Side Effects | Up to 1 year
  • Change in erectile function measured by the IIEF-15 questionnaire
Continence side effect | Up to 1 year
  • Number of patients with urinary incontinence as determined by the UCLA-EPIC urinary continence questionnaire
Rectal side effects | Up to 1 year
  • Number of patients with grade I-II-III type rectal toxicity
Cancer Control | Six months
  Number of patients having residual prostate cancer at 6 months biopsy

OTHER OUTCOMES:
Role of follow-up MRI | Six months
  • Assessment of postoperative MRI value in predicting residual prostate cancer using biopsy as a reference test
Anxiety | Up to 1 year
  • Change in anxiety levels as measured by significant change in the Memorial Anxiety Scale for Prostate Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Hashim U Ahmed, PhD, Principal Investigator — UCLH; Mark Emberton, Professor, Principal Investigator — UCLH
Locations (1):
- University College London Hospitals, London, United Kingdom